CLINICAL TRIAL: NCT03337594
Title: Gadolinium Retention in Human Bone Tissue in Pediatric Patients: a Comparison of Dotarem Versus MultiHance MRI Contrast Agents
Brief Title: Gadolinium Retention in Human Bone Tissue in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Donna Roberts (Other)
Collaborators: National Institute of Standards and Technology (Unknown)
Responsible Party: Sponsor-Investigator, Donna Roberts, Professor, Radiology and Radiological Science Department, Medical University of South Carolina
Organization: Medical University of South Carolina (Other)
Other Study IDs: Pro00048639
Record Dates: First submitted 2017-11-06; First posted 2017-11-09 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-07

CONDITIONS: Gadolinium; MultiHance; Dotarem; Magnetic Resonance Imaging; Gadolinium Retention
Keywords: Gadolinium; MultiHance; Dotarem; Contrast agents; Magnetic Resonance Imaging; Gadolinium retention; Pediatric; Bone
MeSH Terms: interventions — gadoterate meglumine; gadobenic acid; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bone and possibly skin tissue that are removed for routine care during the pediatric cardiothoracic surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Control: Pediatric patients who have not been exposed to gadolinium-based contrast agent administration and who require cardiac surgery as part of their standard clinical treatment.
  Interventions: Procedure: Surgery
- Dotarem: Pediatric patients who have undergone routine contrast-enhanced MRI using only Dotarem contrast agent for clinical purposes and who require cardiac surgery as part of their standard clinical treatment.
  Interventions: Drug: Pre-operative MRI with Dotarem; Procedure: Surgery
- MultiHance: Pediatric patients who have undergone routine contrast-enhanced MRI using only MultiHance contrast agent for clinical purposes and who require cardiac surgery as part of their standard clinical treatment.
  Interventions: Drug: Pre-operative MRI with MultiHance; Procedure: Surgery

INTERVENTIONS:
Drug: Pre-operative MRI with Dotarem — Dotarem® (gadoterate meglumine - Guerbet)
  Other Names: gadoterate meglumine
  Groups: Dotarem
Drug: Pre-operative MRI with MultiHance — MultiHance® (gadobenate dimeglumine - Bracco)
  Other Names: gadobenate dimeglumine
  Groups: MultiHance
Procedure: Surgery — Cardiac surgery

SUMMARY:
The purpose of this study is to compare contrast agents, Dotarem or MultiHance. The study will test to see how much of these two contrast agents are deposited in the bones or tissues of pediatric patients. The patients receiving contrast will then be compared against pediatric patients who have not received any contrast prior to cardiac surgeries.

DETAILED DESCRIPTION:
When injected into the body, gadolinium contrast medium makes certain tissues, abnormalities or disease processes more clearly visible on a magnetic resonance imaging (MRI) scans and therefore gadolinium based contrast agents (GBCAs) are widely used in medical imaging. Recently, new evidence suggests that following GBCA administration, gadolinium can be deposited in body tissues even in the presence of normal renal function. Therefore, it is essential to ensure that significant accumulation of free Gd3+ is not occurring in the bones of children undergoing clinical contrasted MRI scans. This is particularly important for those pediatric patients who will undergo multiple repeated MRI exams throughout their lifetime and thereby be exposed to a large cumulative dose of gadolinium contrast. As the differences in stability between the various GBCAs may be a factor in gadolinium exposure, the primary objective of this study is to assess gadolinium deposition in the bones of pediatric patients in two patient groups: 1. patients who received IV administration of gadolinium contrast agent (Dotarem) and 2. patients who received IV administration of gadolinium contrast agent (MultiHance).

Once acquired the samples will be analyzed at an off-site facility, National Institute of Standards and Technology (NIST), using standardized equipment which has been certified for measuring gadolinium concentration in contrast agent samples. A signed agreement for the transfer of non-proprietary biological material between MUSC and NIST covers the transfer of the samples.

ELIGIBILITY:
Inclusion Criteria:

* Female or male pediatric patient (patients aged newborn to 18 years old at the time of the MRI scan).
* Patients who require cardiac surgery for clinical purposes and meet one of the following three criteria:

  1. Patients who have undergone a routine contrast-enhanced MRI using MultiHance contrast agent only for clinical purposes.
  2. Patients who have undergone a routine contrast-enhanced MRI using Dotarem contrast agent only for clinical purposes.
  3. Patients who have not been exposed to gadolinium-based contrast agent administration

Exclusion Criteria:

* Patient with abnormal renal function (defined as eGFR MDRD<30 ml/min/1.73m2).
* Patient previously exposed to any other type of MRI gadolinium based contrast agent either at MUSC or at an outside facility
* Pregnant or breast feeding female patient
* Patient with a contraindication to MRI (e.g., pacemaker, aneurysm clip, severe claustrophobia, infusion pumps, cochlear implants metallic or others according to standard practice at MUSC).

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All subjects, newborn to 18 years, scheduled for a prospective clinically indicated, contrast-enhanced, cardiac MRI will potentially be eligible for inclusion into the study. Potential subjects will be identified via pediatric cardiology, pediatric cardiothoracic surgery, or clinical schedules and consultation with attending physicians according to satisfaction of the inclusion and exclusion criteria listed above.
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
To determine the gadolinium concentration present in bone tissue in pediatric patients following a standard of care MRI with MultiHance, Dotarem, or without any exposure to contrast. | July 2017 to October 2022
  To determine the gadolinium concentration present in sternum and rib bone tissue in 2 groups of pediatric patients requiring cardiac surgery as part of their standard clinical treatment: (1) patients who had undergone the administration of a standard clinical dose of a linear GBCA (0.1 mmol/kg IV MultiHance), and (2) patients who had undergone the administration of a standard clinical dose of a macrocyclic GBCA (0.1 mmol/kg IV Dotarem). As a control, gadolinium concentration present in sternum bone tissue will also be determined in patients who had not been exposed to GBCA administration prior to surgery.

SECONDARY OUTCOMES:
Asses the number of exposures to contrast agent as a potential confounder. | July 2017 to October 2022
  Number of exposures to contrast agent is a potential confounder. Thus we will perform linear regression, with concentration as the outcome, and both type of contrast agent (i.e. group) and number of doses as independent variables. Although the sample size is small, we may consider evaluating an interaction between type of contrast and number of doses as an exploratory analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Donna R Roberts, M.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hesselink JR, Press GA. MR contrast enhancement of intracranial lesions with Gd-DTPA. Radiol Clin North Am. 1988 Jul;26(4):873-87. PMID 3289078
- [Background] Hesselink JR, Healy ME, Press GA, Brahme FJ. Benefits of Gd-DTPA for MR imaging of intracranial abnormalities. J Comput Assist Tomogr. 1988 Mar-Apr;12(2):266-74. doi: 10.1097/00004728-198803000-00015. PMID 3351041
- [Background] Sherry AD, Caravan P, Lenkinski RE. Primer on gadolinium chemistry. J Magn Reson Imaging. 2009 Dec;30(6):1240-8. doi: 10.1002/jmri.21966. PMID 19938036
- [Background] Bellin MF, Van Der Molen AJ. Extracellular gadolinium-based contrast media: an overview. Eur J Radiol. 2008 May;66(2):160-7. doi: 10.1016/j.ejrad.2008.01.023. Epub 2008 Mar 20. PMID 18358659
- [Background] Hasebroock KM, Serkova NJ. Toxicity of MRI and CT contrast agents. Expert Opin Drug Metab Toxicol. 2009 Apr;5(4):403-16. doi: 10.1517/17425250902873796. PMID 19368492
- [Background] Darrah TH, Prutsman-Pfeiffer JJ, Poreda RJ, Ellen Campbell M, Hauschka PV, Hannigan RE. Incorporation of excess gadolinium into human bone from medical contrast agents. Metallomics. 2009 Nov;1(6):479-88. doi: 10.1039/b905145g. Epub 2009 Sep 16. PMID 21305156
- [Background] White GW, Gibby WA, Tweedle MF. Comparison of Gd(DTPA-BMA) (Omniscan) versus Gd(HP-DO3A) (ProHance) relative to gadolinium retention in human bone tissue by inductively coupled plasma mass spectroscopy. Invest Radiol. 2006 Mar;41(3):272-8. doi: 10.1097/01.rli.0000186569.32408.95. PMID 16481910
- [Background] Port M, Idee JM, Medina C, Robic C, Sabatou M, Corot C. Efficiency, thermodynamic and kinetic stability of marketed gadolinium chelates and their possible clinical consequences: a critical review. Biometals. 2008 Aug;21(4):469-90. doi: 10.1007/s10534-008-9135-x. Epub 2008 Mar 15. PMID 18344005
- [Background] Morcos SK. Extracellular gadolinium contrast agents: differences in stability. Eur J Radiol. 2008 May;66(2):175-9. doi: 10.1016/j.ejrad.2008.01.025. Epub 2008 Mar 14. PMID 18343072
- See also: Link to contact Dr. Roberts — http://academicdepartments.musc.edu/facultydirectory/Roberts-Donna
- See also: NIST: National Institute of Standards and Technology — https://www.nist.gov/